CLINICAL TRIAL: NCT04062240
Title: Bispectral Index: A Comparison of Bifrontal Montage Agreement
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew J. Ritter, Principal Investigator, Mayo Clinic
Other Study IDs: 19-000568
Record Dates: First submitted 2019-08-16; First posted 2019-08-20 (Actual); Results first posted 2023-02-21 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2022-05

CONDITIONS: Surgery; Bispectral Index
Keywords: BIS; Bispectral Index; Paralysis
MeSH Terms: conditions — Paralysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Additional BIS sensor: Many providers caring for cardiovascular surgical patients utilizes BIS monitoring to gauge depth of anesthesia. The current practice involves placement of the BIS sensor on the patient's forehead per the manufacturer's recommendation on arrival to the operating room. The intervention in this study will add an additional BIS sensor to the patient's forehead. After syncing the two monitors for time, and ensuring appropriate skin contact and signal quality of both sensors, BIS monitoring will commence. BIS readings will be available every 12 seconds during the duration of the study, yielding up to 240 points of comparison per enrolled patient.
  Interventions: Device: BIS sensor

INTERVENTIONS:
Device: BIS sensor — BIS sensors will be labeled L and R. The degree of variability between the concurrent use of the sensors will be assessed .

SUMMARY:
The researchers are trying to compare the results of two sensors when recorded simultaneously on opposite sides of the forehead.

DETAILED DESCRIPTION:
Bispectral Index (BIS) monitors are FDA approved to gauge depth of sedation by analyzing segments of electroencephalogram (EEG) waves. The BIS monitor utilizes a proprietary algorithm to process the EEG information second by second, and outputs a number (0-100) that corresponds with a patient's level of consciousness. A level of 0 indicates no EEG activity; a level of 100 indicates awake EEG activity. Several studies demonstrated that BIS monitors may not be useful in paralyzed patients, as patients who were paralyzed and not sedated unexpectedly showed a large decrease in their BIS values following administration paralytic medications. Vivien et al found BIS values dropped an average of 24 points in already sedated patients when the patients were given paralytics. In the same year, Messner and colleagues paralyzed non-sedated volunteers and found a dramatic drop in BIS values until paralysis wore off or was reversed. Schuller et al repeated the Messner experiment and found similar results with 18 of 20 non-sedated volunteer's BIS values dropping to levels expected of patients who were sedated. These results suggest that BIS monitors are integrating electromyography (EMG) data into its algorithm to derive a BIS value. Our hypothesis is that a BIS monitor commenced after paralysis, thereby lacking exposure to any "awake" EMG activity, will result in a cleaner data set and more accurate representation of a patient's level of sedation. Studying in this manner will require the subject to wear two BIS sensors in a frontal montage. The manufacturer of the sensors gives no guidance as to which side of the forehead an individual sensor is placed, and no studies demonstrate BIS validity with the use of concurrent sensors. The purpose of the present investigation is to assess the measurement difference and variability associated with use of concurrent bifrontal BIS sensors. The data obtained will be used as a framework for a future study related to the use of paralytics and BIS monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient having elective cardiac surgery

Exclusion Criteria:

1. Patient refusal.
2. Pediatric patients.
3. Emergency procedure.
4. Patients with known or suspected carotid or cerebrovascular disease.
5. Patients with prior stroke.
6. Skin condition or anatomy preventing proper sensor placement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients undergoing elective cardiac surgery, for whom BIS monitoring will be used.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ritter, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Messner M, Beese U, Romstock J, Dinkel M, Tschaikowsky K. The bispectral index declines during neuromuscular block in fully awake persons. Anesth Analg. 2003 Aug;97(2):488-491. doi: 10.1213/01.ANE.0000072741.78244.C0. PMID 12873942
- [Result] Schuller PJ, Newell S, Strickland PA, Barry JJ. Response of bispectral index to neuromuscular block in awake volunteers. Br J Anaesth. 2015 Jul;115 Suppl 1:i95-i103. doi: 10.1093/bja/aev072. PMID 26174308
- [Result] Vivien B, Di Maria S, Ouattara A, Langeron O, Coriat P, Riou B. Overestimation of Bispectral Index in sedated intensive care unit patients revealed by administration of muscle relaxant. Anesthesiology. 2003 Jul;99(1):9-17. doi: 10.1097/00000542-200307000-00006. PMID 12826836
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Additional Bispectral Index (BIS) Sensor: Many providers caring for cardiovascular surgical patients utilizes BIS monitoring to gauge depth of anesthesia. The current practice involves placement of the BIS sensor on the patient's forehead per the manufacturer's recommendation on arrival to the operating room. The intervention in this study will add an additional BIS sensor to the patient's forehead. After syncing the two monitors for time, and ensuring appropriate skin contact and signal quality of both sensors, BIS monitoring will commence. BIS readings will be available every 12 seconds during the duration of the study, yielding up to 240 points of comparison per enrolled patient.
  BIS sensor: BIS sensors will be labeled L and R. The degree of variability between the concurrent use of the sensors will be assessed .
Period: Overall Study
Arm/Group | Additional Bispectral Index (BIS) Sensor
Started | 15
Completed | 14
Not Completed | 1
Not completed — equipment malfunction | 1

BASELINE CHARACTERISTICS:
Arm/Group | Additional BIS Sensor
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: BIS Montage
Description: Degree of variability between the values produced by the BIS sensors in a bifrontal montage when monitored simultaneously by use of a Bland-Altmann plot. The average value of each timed pair was plotted against the difference between the pairs.
  The BIS monitor outputs data on a scale of 0-100 in arbitrary units; 0 = an isoelectric state on EEG, 100 = fully awake patient. BIS values of 40-60 are thought to reduce the chance of patient recall during general anesthesia.
  For the purpose of this study, a smaller confidence interval is better as it indicates a higher level of agreement between the two BIS sensors.
Time Frame: 10 minutes where both sensors are recording concurrently
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Additional BIS Sensor
Number analyzed (Participants) | 14
units on a scale | 0.01 [-8.01 to 8.03]

2. Secondary Outcome: Ketamine
Description: Degree to which Ketamine may influence BIS values
Time Frame: 10 minutes where both sensors are recording concurrently
Population: Due to the inconsistent usage and dosages of ketamine administered to the study population, no data was collected to examine this secondary measure.
Arm/Group | Additional BIS Sensor
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for approximately a 10 minute period in the operating room on all participants.
Arm/Group | Additional BIS Sensor
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-19): https://cdn.clinicaltrials.gov/large-docs/40/NCT04062240/Prot_SAP_000.pdf